CLINICAL TRIAL: NCT03285321
Title: Phase II Study of Consolidation Immunotherapy With Nivolumab and Ipilimumab or Nivolumab Alone Following Concurrent Chemoradiotherapy for Unresectable Stage IIIA/IIIB Non-small Cell Lung Cancer (NSCLC): BTCRC-LUN16-081
Brief Title: Unresectable Stage IIIA/IIIB Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Greg Durm, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry); Big Ten Cancer Research Consortium (Other)
Responsible Party: Sponsor-Investigator, Greg Durm, MD, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-LUN16-081
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Nivolumab; Ipilimumab; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Masking Description: Open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Nivolumab 480mg IV every 4 weeks for up to 6 cycles
  Interventions: Drug: Nivolumab
- Arm 2 (Experimental): Nivolumab 240mg IV every 2 weeks PLUS Ipilimumab 1mg/kg IV every 6 weeks for up to 4 cycles (12 doses Nivolumab and 4 doses of Ipilimumab)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — 480mg
  Other Names: OPDIVO
  Arms: Arm 1
Drug: Nivolumab — 240mg
  Other Names: OPDIVO
  Arms: Arm 2
Drug: Ipilimumab — 1mg/kg
  Other Names: Yervoy
  Arms: Arm 2

SUMMARY:
This study is an open label, multicenter, randomized phase II trial of consolidation immunotherapy with either nivolumab alone or the combination of nivolumab and ipilimumab following concurrent chemoradiation in patients with unresectable stage III NSCLC.

DETAILED DESCRIPTION:
Patients with unresectable stage IIIA or IIIB NSCLC (unresectable as defined by treating physician) will be treated outside this study with concurrent chemoradiation with one of three chemotherapy regimens (cisplatin/etoposide, cisplatin/pemetrexed, or weekly carboplatin/paclitaxel) in addition to standard dose radiation (dosing can range from 59.4 Gy to 66.6 Gy). If repeat imaging between 28-56 days following completion of chemoradiation shows no progressive or metastatic disease, the patients will be eligible for enrollment on the study.

Randomization and Stratification:

At the time of enrollment, patients will be randomized in a 1:1 fashion to receive either nivolumab 480mg IV every 4 weeks or the combination of nivolumab 3mg/kg IV every 2 weeks with ipilimumab 1mg/kg IV every 6 weeks. Consolidation immunotherapy will be continued until progression or unacceptable toxicity for up to a total of 24 weeks.

Subjects will be stratified by stage (IIIA vs. IIIB) and histology (squamous vs. non-squamous).

Dose Calculations:

Arm 1: The dose of nivolumab will be a fixed dose (not based on subject's weight) at 480mg.

Arm 2: The dose of nivolumab will be weight-based at 3mg/kg. The dose of ipilimumab will be weight-based at 1mg/kg.

Nivolumab Alone (Arm 1):

Arm 1: Nivolumab Administration:

Nivolumab 480 mg will be administered as a 60 minute IV infusion on Day 1 of each 28 day cycle. Sites should make every effort to target infusion timing to be as close to 60 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -five minutes and +10 minutes is permitted (i.e., infusion time is 60 minutes: -5 min/+10 min). Treatment will continue for up to 6 cycles, in the absence of prohibitive toxicities or disease progression.

Nivolumab Plus Ipilimumab (Arm 2):

Arm 2: Nivolumb Administration:

Nivolumab 3mg/kg will be administered as a 60 minute IV infusion on Day 1, 15, and 29 of each 42 day cycle. Nivolumab should not be given any earlier than 12 days from the previous dose. Sites should make every effort to target infusion timing to be as close to 60 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -five minutes and +10 minutes is permitted (i.e., infusion time is 60 minutes: -5 min/+10 min). Treatment will continue for up to 4 cycles, in the absence of prohibitive toxicities or disease progression.

Arm 2: Ipilimumab Administration:

Ipilimumab 1mg/kg will be administered as a 90 minute IV infusion on Day 1 of each 42 day cycle. Sites should make every effort to target infusion timing to be as close to 90 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -five minutes and +10 minutes is permitted (i.e., infusion time is 60 minutes: -5 min/+10 min). Treatment will continue for up to 4 cycles, in the absence of prohibitive toxicities or disease progression.

On day 1 of cycle 1, nivolumab will be given first, followed by 30 minutes of monitoring, and then ipilimumab given second, followed by 30 minutes of monitoring. If the subject does not have an infusion reaction during the first cycle, the post-ipilimumab monitoring may be discontinued for subsequent cycles at the discretion of the treating physician. Day 1 monitoring between the nivolumab/ipilimumab infusions will continue throughout all 4 cycles. Post nivolumab monitoring on days 15 and 29 is not mandatory and should follow the guidelines of the local infusion center.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0 or 1 within 14 days prior to registration.
* Histological or cytological confirmation of NSCLC. A pathology report confirming the diagnosis of NSCLC must be obtained and reviewed by the treating physician prior to registration to study.
* Must have unresectable or inoperable stage IIIA or IIIB disease according to the 7th edition IASLC stage classification for lung cancer. Subjects must be considered unresectable or inoperable based on the judgment of the treating physician.
* Subjects must have completed concurrent chemoradiation with a platinum doublet and a dose of radiation ranging from 59.4-66.6 Gy. Subjects must have stable disease or disease response as evidenced on CT or PET scan evaluation. For those eligible, protocol therapy should begin within 56 days of completing chemoradiation OR Subjects must have completed up to 2 cycles of consolidation therapy started within 56 days of completion of radiation. After completion of consolidation chemotherapy, subjects must have stable disease or disease response as evidenced by CT or PET scan evaluation. For those eligible, protocol therapy should begin within 56 days after the last cycle of chemotherapy.
* Prior cancer treatment must be completed between 1-56 days prior to registration and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤Grade 1 or baseline.
* Demonstrate adequate organ function, all screening labs to be obtained within 14 days prior to registration:

Hematological:

* Absolute Neutrophil Count (ANC) ≥ 1.5 K/mm^3
* Hemoglobin (Hgb) ≥ 9 g/dL
* Platelets ≥100,000/mcl

Renal:

* Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ 1.5 x upper limit of normal (ULN) OR ≥ 60 mL/min for subjects with creatinine levels >1.5 x institutional ULN

Hepatic:

* Bilirubin ≤ 1.5 × ULN OR Direct bilirubin of ≤ ULN for subjects with total bilirubin levels of >1.5x ULN
* Aspartate aminotransferase (AST) ≤ 2.5 × ULN
* Alanine aminotransferase (ALT) ≤ 2.5 × ULN

Coagulation:

* International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT/INR/PTT is within therapeutic range of intended use of anticoagulants

  * Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to registration. NOTE: Women are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are post-menopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 62 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL to be considered post-menopausal.
  * Women of childbearing potential must be willing to abstain from heterosexual activity or use an effective method of contraception from the time of informed consent until 23 weeks after treatment discontinuation.
  * Men who are sexually active with women of childbearing potential (WOCBP) must use any contraceptive method with a failure rate of less than 1% per year. Men receiving study drug and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product.
  * As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 23 weeks (female) or 31 weeks (male) after the last dose of trial treatment.
* Active central nervous system (CNS) metastases. Subjects must undergo a head computed tomography (CT) scan or brain MRI within 28 days prior to registration for protocol therapy to exclude brain metastases if symptomatic or without prior brain imaging.
* Treatment with any investigational agent within 28 days prior to registration for protocol therapy.
* Prior chemotherapy, adjuvant therapy, or radiotherapy for lung cancer other than standard concurrent chemoradiation or up to 2 cycles of consolidation.
* Prior therapy with a PD-1, PD-L1, PD-L2 or CTLA-4 inhibitor or a lung cancer-specific vaccine therapy.
* Presence of metastatic disease (stage IV NSCLC) is not allowed. Subjects must be evaluated with a CT or PET scan prior to registration for protocol therapy to exclude metastatic disease.
* Active second cancers.
* Evidence of active autoimmune disease requiring systemic treatment within the past 90 days or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
* Interstitial lung disease or history of pneumonitis requiring treatment with corticosteroids.
* Diagnosis of immunodeficiency or is receiving chronic systemic corticosteroid therapy or other immunosuppressive therapy (excludes inhaled corticosteroids) within 7 days of first dose of study drug.
* History of psychiatric illness or social situations that would limit compliance with study requirements.
* Clinically active infection as judged by the site investigator (≥ Grade 2 by CTCAE v4).
* History of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the site investigator.
* Has a known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to nivolumab, ipilimumab, or any of their excipients.
* Has received a live vaccine within 30 days prior to planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2024-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Durm, M.D., Study Chair — Indiana University Health Simon Cancer Center
Locations (12):
- United States (12):
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - Johns Hopkins Sidney Kimmel Comprehensive, Baltimore, Maryland
  - Karmanos Cancer Center (Wayne State University), Detroit, Michigan
  - Michigan State University, Lansing, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Nivolumab: Nivolumab 480mg IV every 4 weeks for up to 6 cycles
  Nivolumab: 480mg
- Arm 2: Nivolumab Plus Ipilimumab: Nivolumab 240mg IV every 2 weeks PLUS Ipilimumab 1mg/kg IV every 6 weeks for up to 4 cycles (12 doses Nivolumab and 4 doses of Ipilimumab)
  Nivolumab: 240mg
  Ipilimumab: 1mg/kg
Period: Overall Study
Arm/Group | Arm 1: Nivolumab | Arm 2: Nivolumab Plus Ipilimumab
Started | 54 | 51
Completed | 54 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Nivolumab | Arm 2: Nivolumab Plus Ipilimumab | Total
Number analyzed (Participants) | 54 | 51 | 105
Age, Continuous [Median (Full Range); unit: years] | 65 [44 to 82] | 63 [41 to 83] | 64 [41 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 22 | 52
  Male | 24 | 29 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 16 | 26
  White | 42 | 30 | 72
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 54 | 51 | 105
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction, 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, and 5=Dead.
  Participants
    ECOG = 0 | 18 | 27 | 45
    ECOG = 1 | 36 | 24 | 60

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) at 18-month
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  PFS is defined as the time from randomization until the criteria for disease progression is met as defined by RECIST 1.1 or death as a result of any cause.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Nivolumab | Arm 2: Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 54 | 51
Percentage of participants | 65.5 [49.8 to 77.3] | 66.3 [56.3 to 74.5]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization until death from any cause.
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Nivolumab | Arm 2: Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 54 | 51
Months | 32 [32 to NA] — Not enough events occur to calculate the upper 95% confidence interval. | NA [30.9 to NA] — Not enough events occur to calculate the median and upper 95% confidence interval.

3. Secondary Outcome: Time to Metastatic Disease (TTMD) at 36 Month
Description: TTMD is defined as the time from randomization until evidence of disease outside of the radiated field. The estimate of TTMD at 36 month with 95% confidence interval are reported in the outcome measure data.
Time Frame: 36 Months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: Nivolumab | Arm 2: Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 54 | 51
Percentage of participants | 79.7 [61 to 90.1] | 77.5 [58.2 to 88.7]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be assessed to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nivolumab | Arm 2: Nivolumab Plus Ipilimumab
Number analyzed (Participants) | 54 | 51
Participants | 54 | 51

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 4 Years. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 12 months.
Arm/Group | Arm 1: Nivolumab | Arm 2: Nivolumab Plus Ipilimumab
All-Cause Mortality (participants affected / at risk) | 14/54 | 15/51
Serious Adverse Events (participants affected / at risk) | 10/54 | 21/51
Other Adverse Events (participants affected / at risk) | 52/54 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Nivolumab (N=54) | Arm 2: Nivolumab Plus Ipilimumab (N=51)
ATRIAL FIBRILLATION (CARDIAC DISORDERS) | 1 (1) | 0 (0)
CHEST PAIN - CARDIAC (CARDIAC DISORDERS) | 1 (1) | 0 (0)
DYSPNEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 3 (5)
HEART FAILURE (CARDIAC DISORDERS) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (INFECTIONS AND INFESTATIONS) | 1 (1) | 1 (1)
LUNG INFECTION (INFECTIONS AND INFESTATIONS) | 3 (3) | 3 (4)
NON-CARDIAC CHEST PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1) | 0 (0)
PNEUMONITIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 5 (5) | 9 (10)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0)
SEPSIS (INFECTIONS AND INFESTATIONS) | 2 (2) | 0 (0)
SINUS TACHYCARDIA (CARDIAC DISORDERS) | 1 (1) | 0 (0)
THROMBOEMBOLIC EVENT (VASCULAR DISORDERS) | 1 (1) | 2 (2)
URTICARIA (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1) | 0 (0)
BRONCHOPULMONARY HEMORRHAGE (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
CARDIAC ARREST (CARDIAC DISORDERS) | 0 (0) | 1 (1)
COGNITIVE DISTURBANCE (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
COLITIS (GASTROINTESTINAL DISORDERS) | 0 (0) | 2 (2)
DEHYDRATION (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 1 (1)
FEVER (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (2)
HYPERGLYCEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 1 (1)
HYPONATREMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 1 (1)
HYPOXIA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 2 (2)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (IMMUNE SYSTEM DISORDERS) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (CARDIAC DISORDERS) | 0 (0) | 1 (1)
PANCREATITIS (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
PLEURAL EFFUSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 2 (2)
RESPIRATORY FAILURE (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Nivolumab (N=54) | Arm 2: Nivolumab Plus Ipilimumab (N=51)
ABDOMINAL PAIN (GASTROINTESTINAL DISORDERS) | 1 (1) | 4 (4)
ACUTE CORONARY SYNDROME (CARDIAC DISORDERS) | 1 (1) | 0 (0)
AGITATION (PSYCHIATRIC DISORDERS) | 1 (1) | 1 (3)
ALANINE AMINOTRANSFERASE INCREASED (INVESTIGATIONS) | 3 (3) | 2 (2)
ALKALINE PHOSPHATASE INCREASED (INVESTIGATIONS) | 2 (3) | 4 (10)
ALLERGIC RHINITIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 (2) | 6 (7)
ALOPECIA (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1) | 0 (0)
ANEMIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 6 (6) | 13 (18)
ANKLE FRACTURE (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1) | 0 (0)
ANOREXIA (METABOLISM AND NUTRITION DISORDERS) | 6 (7) | 8 (12)
ANXIETY (PSYCHIATRIC DISORDERS) | 4 (4) | 2 (3)
ARTHRALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 3 (4) | 7 (13)
ARTHRITIS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 2 (3) | 3 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (INVESTIGATIONS) | 3 (4) | 4 (7)
ATRIAL FIBRILLATION (CARDIAC DISORDERS) | 1 (1) | 0 (0)
BACK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 8 (13) | 7 (9)
BLADDER INFECTION (INFECTIONS AND INFESTATIONS) | 2 (2) | 0 (0)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 3 (3) | 3 (5)
BLURRED VISION (EYE DISORDERS) | 3 (3) | 2 (2)
BRONCHIAL INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1) | 1 (1)
BRONCHOSPASM (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0)
BRUISING (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1) | 1 (1)
BULLOUS DERMATITIS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1) | 0 (0)
CARDIAC DISORDERS - OTHER, SPECIFY (CARDIAC DISORDERS) | 2 (2) | 1 (2)
CHEST WALL PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 3 (3) | 0 (0)
CHILLS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 2 (3) | 4 (6)
CHOLESTEROL HIGH (INVESTIGATIONS) | 2 (2) | 1 (1)
CONFUSION (PSYCHIATRIC DISORDERS) | 1 (1) | 2 (3)
CONSTIPATION (GASTROINTESTINAL DISORDERS) | 5 (5) | 7 (8)
COUGH (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 16 (16) | 24 (29)
CREATININE INCREASED (INVESTIGATIONS) | 6 (11) | 5 (5)
DEHYDRATION (METABOLISM AND NUTRITION DISORDERS) | 4 (4) | 3 (4)
DENTAL CARIES (GASTROINTESTINAL DISORDERS) | 1 (1) | 0 (0)
DEPRESSION (PSYCHIATRIC DISORDERS) | 3 (4) | 1 (1)
DIARRHEA (GASTROINTESTINAL DISORDERS) | 9 (13) | 16 (24)
DIZZINESS (NERVOUS SYSTEM DISORDERS) | 10 (11) | 10 (11)
DRY MOUTH (GASTROINTESTINAL DISORDERS) | 4 (4) | 3 (5)
DRY SKIN (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 2 (2) | 2 (2)
DYSGEUSIA (NERVOUS SYSTEM DISORDERS) | 1 (1) | 3 (6)
DYSPHAGIA (GASTROINTESTINAL DISORDERS) | 4 (4) | 2 (2)
DYSPHASIA (NERVOUS SYSTEM DISORDERS) | 1 (1) | 0 (0)
DYSPNEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 18 (23) | 24 (46)
EAR PAIN (EAR AND LABYRINTH DISORDERS) | 1 (1) | 0 (0)
EDEMA LIMBS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 5 (5) | 7 (9)
ENDOCRINE DISORDERS - OTHER, SPECIFY (ENDOCRINE DISORDERS) | 3 (4) | 1 (1)
ERECTILE DYSFUNCTION (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 1 (1) | 0 (0)
ERYTHEMA MULTIFORME (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (2) | 1 (1)
ESOPHAGEAL ULCER (GASTROINTESTINAL DISORDERS) | 1 (1) | 0 (0)
ESOPHAGITIS (GASTROINTESTINAL DISORDERS) | 2 (2) | 0 (0)
EYE DISORDERS - OTHER, SPECIFY (EYE DISORDERS) | 1 (1) | 0 (0)
FALL (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 3 (3) | 3 (3)
FATIGUE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 22 (35) | 25 (40)
FEVER (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 5 (10) | 6 (7)
FLANK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 2 (2)
FLATULENCE (GASTROINTESTINAL DISORDERS) | 1 (1) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEASE (GASTROINTESTINAL DISORDERS) | 2 (2) | 2 (3)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 4 (5) | 8 (14)
GUM INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1) | 0 (0)
HEADACHE (NERVOUS SYSTEM DISORDERS) | 12 (12) | 16 (18)
HEARING IMPAIRED (EAR AND LABYRINTH DISORDERS) | 1 (2) | 1 (1)
HEMATURIA (RENAL AND URINARY DISORDERS) | 1 (1) | 0 (0)
HOARSENESS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 (2) | 2 (4)
HYPERGLYCEMIA (METABOLISM AND NUTRITION DISORDERS) | 2 (2) | 3 (3)
HYPERHIDROSIS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1) | 3 (5)
HYPERKALEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (3) | 1 (1)
HYPERTENSION (VASCULAR DISORDERS) | 3 (4) | 1 (1)
HYPERTHYROIDISM (ENDOCRINE DISORDERS) | 3 (3) | 1 (1)
HYPOKALEMIA (METABOLISM AND NUTRITION DISORDERS) | 7 (11) | 9 (17)
HYPOMAGNESEMIA (METABOLISM AND NUTRITION DISORDERS) | 9 (10) | 6 (11)
HYPONATREMIA (METABOLISM AND NUTRITION DISORDERS) | 4 (5) | 5 (12)
HYPOPHOSPHATEMIA (METABOLISM AND NUTRITION DISORDERS) | 2 (2) | 3 (5)
HYPOTENSION (VASCULAR DISORDERS) | 1 (1) | 4 (5)
HYPOTHYROIDISM (ENDOCRINE DISORDERS) | 11 (15) | 9 (14)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (INFECTIONS AND INFESTATIONS) | 1 (1) | 2 (3)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1) | 1 (1)
INSOMNIA (PSYCHIATRIC DISORDERS) | 4 (4) | 10 (12)
JOINT EFFUSION (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 0 (0)
LARYNGITIS (INFECTIONS AND INFESTATIONS) | 1 (1) | 1 (1)
LIBIDO DECREASED (PSYCHIATRIC DISORDERS) | 1 (1) | 0 (0)
LUNG INFECTION (INFECTIONS AND INFESTATIONS) | 9 (14) | 10 (15)
LYMPHOCYTE COUNT DECREASED (INVESTIGATIONS) | 1 (1) | 2 (6)
MEMORY IMPAIRMENT (NERVOUS SYSTEM DISORDERS) | 1 (1) | 0 (0)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (METABOLISM AND NUTRITION DISORDERS) | 3 (3) | 0 (0)
MUSCLE WEAKNESS LOWER LIMB (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 2 (2) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 5 (8) | 6 (8)
MYALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 5 (7) | 3 (5)
MYOSITIS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 1 (3)
NASAL CONGESTION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 (2) | 7 (11)
NAUSEA (GASTROINTESTINAL DISORDERS) | 13 (13) | 15 (25)
NECK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 1 (1)
NEUTROPHIL COUNT DECREASED (INVESTIGATIONS) | 1 (1) | 1 (1)
NON-CARDIAC CHEST PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 9 (11) | 5 (8)
ORAL PAIN (GASTROINTESTINAL DISORDERS) | 1 (1) | 0 (0)
PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 10 (11) | 11 (15)
PAIN IN EXTREMITY (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 4 (6) | 7 (10)
PERIPHERAL SENSORY NEUROPATHY (NERVOUS SYSTEM DISORDERS) | 6 (7) | 6 (6)
PLEURAL EFFUSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 4 (6)
PNEUMONITIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 10 (22) | 15 (25)
PNEUMOTHORAX (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 6 (8) | 6 (9)
PRURITUS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 8 (10) | 14 (25)
RASH ACNEIFORM (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 10 (18) | 12 (18)
RECTAL HEMORRHAGE (GASTROINTESTINAL DISORDERS) | 1 (1) | 1 (1)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (RENAL AND URINARY DISORDERS) | 1 (1) | 0 (0)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER, SPECIFY (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 7 (8) | 4 (4)
RETINOPATHY (EYE DISORDERS) | 1 (1) | 0 (0)
RHINITIS INFECTIVE (INFECTIONS AND INFESTATIONS) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (CARDIAC DISORDERS) | 2 (2) | 4 (5)
SINUSITIS (INFECTIONS AND INFESTATIONS) | 2 (2) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 7 (8) | 8 (10)
SKIN HYPOPIGMENTATION (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1) | 0 (0)
SKIN INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1) | 2 (2)
SORE THROAT (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 (2) | 0 (0)
SPINAL FRACTURE (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1) | 0 (0)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (SURGICAL AND MEDICAL PROCEDURES) | 2 (2) | 2 (5)
SYNCOPE (NERVOUS SYSTEM DISORDERS) | 1 (1) | 0 (0)
THROMBOEMBOLIC EVENT (VASCULAR DISORDERS) | 4 (7) | 5 (6)
UPPER RESPIRATORY INFECTION (INFECTIONS AND INFESTATIONS) | 3 (3) | 6 (11)
URINARY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1) | 1 (1)
URINARY TRACT PAIN (RENAL AND URINARY DISORDERS) | 1 (1) | 0 (0)
URINARY URGENCY (RENAL AND URINARY DISORDERS) | 1 (1) | 0 (0)
URTICARIA (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1) | 0 (0)
VAGINAL INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1) | 0 (0)
VOMITING (GASTROINTESTINAL DISORDERS) | 3 (3) | 9 (12)
WEIGHT GAIN (INVESTIGATIONS) | 3 (3) | 1 (1)
WEIGHT LOSS (INVESTIGATIONS) | 5 (5) | 9 (13)
WHEEZING (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 (2) | 2 (2)
WHITE BLOOD CELL DECREASED (INVESTIGATIONS) | 2 (2) | 1 (3)
WOUND COMPLICATION (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1) | 0 (0)
ABDOMINAL INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
ADRENAL INSUFFICIENCY (ENDOCRINE DISORDERS) | 0 (0) | 1 (1)
BONE PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 1 (1)
BREAST PAIN (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 0 (0) | 1 (1)
CHEST PAIN - CARDIAC (CARDIAC DISORDERS) | 0 (0) | 1 (1)
COLITIS (GASTROINTESTINAL DISORDERS) | 0 (0) | 2 (2)
CONJUNCTIVITIS (EYE DISORDERS) | 0 (0) | 1 (3)
DYSPEPSIA (GASTROINTESTINAL DISORDERS) | 0 (0) | 2 (3)
EPISTAXIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 4 (4)
FACIAL PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1)
GAIT DISTURBANCE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1)
GASTRITIS (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 3 (5)
HOT FLASHES (VASCULAR DISORDERS) | 0 (0) | 1 (1)
HYPOALBUMINEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 3 (5)
HYPOXIA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (IMMUNE SYSTEM DISORDERS) | 0 (0) | 2 (2)
INVESTIGATIONS - OTHER, SPECIFY (INVESTIGATIONS) | 0 (0) | 2 (3)
LEUKOCYTOSIS (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 0 (0) | 1 (1)
LIPASE INCREASED (INVESTIGATIONS) | 0 (0) | 3 (5)
LOCALIZED EDEMA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 2 (2)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 0 (0) | 2 (2)
PAPULOPUSTULAR RASH (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (2)
PARESTHESIA (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (CARDIAC DISORDERS) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (INVESTIGATIONS) | 0 (0) | 5 (5)
POSTNASAL DRIP (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
PRESYNCOPE (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
PULMONARY FIBROSIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (2)
PULMONARY HYPERTENSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
SEPSIS (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
SERUM AMYLASE INCREASED (INVESTIGATIONS) | 0 (0) | 3 (4)
SINUS PAIN (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
STOMACH PAIN (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (2)
SUPERFICIAL THROMBOPHLEBITIS (VASCULAR DISORDERS) | 0 (0) | 1 (1)
TINNITUS (EAR AND LABYRINTH DISORDERS) | 0 (0) | 1 (1)
TREMOR (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
URINARY FREQUENCY (RENAL AND URINARY DISORDERS) | 0 (0) | 2 (2)
VERTIGO (EAR AND LABYRINTH DISORDERS) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT03285321/Prot_SAP_000.pdf